CLINICAL TRIAL: NCT06599164
Title: Evaluation of Muscular Anthrogenic Inhibition of the Vasto Medialis in Indoor Soccer Players with Anterior Cruciate Ligament (ACL) Injury in Comparison with Non-Injured Players: Observational Cohort Study
Brief Title: Evaluation of Vastus Medialis Muscle Inhibition in Indoor Soccer Players with and Without ACL Injury
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, maria martinez parada, Principal investigador, University of Alcala
Other Study IDs: CEIM/2024/4/095
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anterior Cruciate Ligament Injuries; Knee Injuries
Keywords: Anthrogenic Muscle Inhibition; Soccer; Anterior Cruciate Ligament; Rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- UNINJURED PLAYERS: Players will be evaluated for isometric strength by electromyography, extensor strength, single leg vertical jump test and ultrasound evaluation, all of which will be measured on all players in the preseason, at 4 months and at the end of the season.
  Interventions: Other: Anthrogenic Muscle Inhibition (AMI) Assessment Protocol
- INJURED PLAYERS: As for futsal players with ACL injuries, isometric strength is evaluated in pre-operation, at 4 months and at the end of the soccer year by electromyography, extensor strength, single-leg vertical jump test and ultrasound evaluation.
  Interventions: Other: Anthrogenic Muscle Inhibition (AMI) Assessment Protocol

INTERVENTIONS:
Other: Anthrogenic Muscle Inhibition (AMI) Assessment Protocol — This study involves evaluating Anthrogenic Muscle Inhibition (AMI) of the vastus medialis muscle in futsal players. The intervention includes assessments of muscle strength, AMI using electromyography, ultrasound evaluation, and single-leg vertical jump tests. These evaluations are conducted at different stages throughout the season: pre-season, 4 months in, and at the end of the season. The goal is to compare AMI levels and muscle function between players with ACL injuries and those without.
  Other Names: Vastus Medialis AMI Assessment; Isometric Strength Evaluation Protocol

SUMMARY:
The Anterior Cruciate Ligament (ACL) is vital for knee stability, and ACL injuries in futsal can lead to long-term issues. Reconstruction surgery may be affected by Anthrogenic Muscle Inhibition (AMI), especially in the vastus medialis muscle. This study aims to compare AMI in futsal players with ACL injuries to those without injuries, focusing on measurement techniques, sports performance, muscle strength, and recovery time. The research involves evaluating 54 players (27 injured and 27 non-injured) at various stages of the season using strength tests and imaging.

DETAILED DESCRIPTION:
Introduction: The Anterior Cruciate Ligament (ACL) is crucial for knee stability and represents a major challenge in sports such as futsal. ACL injuries can carry a risk of long-term complications. While reconstruction surgery is a common method for recovery, it can be affected by Anthrogenic Muscle Inhibition (AMI), especially in the vastus medialis. Research on AMI in futsal players will be fundamental to improve rehabilitation, functionality, and reduce the risk of relapse.

Objectives: To analyze the changes in the Anthrogenic Muscular Inhibition of the vastus medialis in futsal players with Anterior Cruciate Ligament Injury compared to non-injured players. The specific objectives include evaluating measurement techniques, assessing the impact on sport quality, assessing muscle strength, and examining recovery time.

Methodology: The present study uses an observational cohort design to evaluate AMI in indoor soccer players at different stages of the soccer season, compared to players who suffer ACL injuries during competition. The sample size is 54 subjects, with 27 in each group. Accounting for a 15% loss, the final sample will be 64 subjects (32 in each group). Players will be evaluated for isometric strength by electromyography, strength in extensors, single leg vertical jump test, and ultrasound evaluation. These measurements will be taken for all players in the pre-season, after 4 months, and at the end of the season. For ACL injuries, evaluations will be conducted pre-operation, 4 months post-operation, and at the end of the soccer year.

Key words: Anthrogenic Muscle Inhibition, soccer, Anterior Cruciate Ligament, Rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years old
* Playing in the Spanish National League (first or second category) or in the Madrid Futsal Federation in PRIMERA RFFM and PREFERENTE.
* Both sexes
* Have been playing futsal for at least 2 years
* Enrolled in the Madrid Health System
* Any language

Exclusion Criteria:

* Operations other than an Anterior Cruciate Ligament injury (Cartilage, Meniscus, Ligaments).
* Injuries to the knee of the contralateral lower limb. (sprains, fracture)
* Muscle injuries or conditions in the affected or contralateral limb for less than 2 months (sprains, tibial periostitis, tendinopathies, tears).
* Any infection must be reported after the intervention and will be excluded from the study.
* Players will not be allowed to play any kind of team sport other than Futsal in an official way during this season.
* Players may not have any cardiovascular or respiratory pathology that would affect the study.
* Players who have already undergone an Anterior Cruciate Ligament rupture in previous years will not be considered.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of futsal players aged 18-45. This includes two groups: (1) players without ACL injuries who serve as a comparison group, and (2) players who have sustained ACL injuries and are undergoing or have undergone ACL reconstruction surgery. The study aims to compare Anthrogenic Muscle Inhibition (AMI) and muscle function between these two groups.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Anthrogenic Muscle Inhibition (AMI) of Vastus Medialis | First 4 weeks (28 days), 4 months (120 days) after the start of the season, and the last 4 months (120 days) of the season. 3 months (90 days) before the operation, 4 months (120 days) after the operation, and the last 4 months (120 days) of the season
  This measure evaluates the level of Anthrogenic Muscle Inhibition (AMI) in the vastus medialis muscle. Assessment Tool: Electromyography and Ultrasound Unit of Measure: Percentage (%)

SECONDARY OUTCOMES:
isometric extension maximum knee with traction | First 4 weeks (28 days), 4 months (120 days) after the start of the season, and the last 4 months (120 days) of the season. 3 months (90 days) before the operation, 4 months (120 days) after the operation, and the last 4 months (120 days) of the season
  this test is used to obtain strength maximum knee extension. For To be able to measure, a cell of strain gauge load fixed to the stretcher where the test will be performed with the knee fixed at 90º. It will be carried out in the two legs, noting which of them is the dominant. Newton (N)
The Single Leg Vertical Jump exercise | First 4 weeks (28 days), 4 months (120 days) after the start of the season, and the last 4 months (120 days) of the season. 3 months (90 days) before the operation, 4 months (120 days) after the operation, and the last 4 months (120 days) of the season
  It is a test used to being able to know the strength, power and capacity that the muscle has where the participant performs a vertical jump with a single leg, in this case it will be 3 times with one and 3 times with the leg contralateral. CM
assessment surface electromyography | First 4 weeks (28 days), 4 months (120 days) after the start of the season, and the last 4 months (120 days) of the season. 3 months (90 days) before the operation, 4 months (120 days) after the operation, and the last 4 months (120 days) of the season
  the function neuromuscular and detect imbalances in muscle activation. HE surface electrodes will be used adhesives to the vastus medialis. To obtain electromyographic tracings patient will perform a contraction maximum isometric 6 seconds duration. microvolts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Booth A, Clarke M, Dooley G, Ghersi D, Moher D, Petticrew M, Stewart L. The nuts and bolts of PROSPERO: an international prospective register of systematic reviews. Syst Rev. 2012 Feb 9;1:2. doi: 10.1186/2046-4053-1-2. PMID 22587842
- [Background] Márquez Arabia WH, Márquez Arabia JJ, Gómez JC. ¿Qué ocurre con las lesiones del ligamento cruzado anterior, su tratamiento, la recuperación de la función y el desarrollo de osteoartritis a largo plazo? ¿Hay espacio para el tratamiento conservador? Revisión de conceptos actuales William. Rev Colomb Ortop y Traumatol. 2017;31(2):75-86
- [Background] Márquez Arabia JJ, Márquez Arabia WH. Lesiones del ligamento cruzado anterior de la rodilla. Iatreia. 2009;22:256-71.
- [Background] Lohmander LS, Englund PM, Dahl LL, Roos EM. The long-term consequence of anterior cruciate ligament and meniscus injuries: osteoarthritis. Am J Sports Med. 2007 Oct;35(10):1756-69. doi: 10.1177/0363546507307396. Epub 2007 Aug 29. PMID 17761605
- [Background] Noyes FR, Barber-Westin SD. Anterior cruciate ligament primary reconstruction: diagnosis, operative techniques, and clinical outcomes. In: Noyes FR, Barber- Westin SD, eds. Noyes&amp;#39; Knee Disorders Surgery, Rehabilitation, Clinical Outcomes. 2nd ed. Philadelphia, PA: Elsevier; 2017:chap 7
- [Background] Calvo Sanz J. Análisis de la inhibición muscular artrogénica del cuádriceps posligamentoplastia del ligamento cruzado anterior de rodilla y su repercusión en la función del aparato extensor [Internet]. TDX (Tesis Doctorals en Xarxa). 2017. Available from: http://www.tdx.cat/handle/10803/432780
- [Background] Williams GN, Barrance PJ, Snyder-Mackler L, Buchanan TS. Altered quadriceps control in people with anterior cruciate ligament deficiency. Med Sci Sports Exerc. 2004 Jul;36(7):1089-97. doi: 10.1249/01.mss.0000131959.20666.11. PMID 15235310
- [Background] Asociacion Española de Artroscopia. Informe sobre el perfil de la cirugía artroscopia en España. Cuadernos de Artroscopia. 2001; 8:10-21
- [Background] Lopez-Segovia M, Vivo Fernandez I, Herrero Carrasco R, Pareja Blanco F. Preseason Injury Characteristics in Spanish Professional Futsal Players: The LNFS Project. J Strength Cond Res. 2022 Jan 1;36(1):232-237. doi: 10.1519/JSC.0000000000003419. PMID 31895285
- [Background] Zamora-Navas P. Evaluacion de la evidencia del tratamiento de las lesiones del ligamento cruzado anterior de la rodilla. Rev Esp Cir Orteoartic. 2005 Jun; 40 (222): 59-66.
- [Background] Lopez-Valenciano A, Ruiz-Perez I, Garcia-Gomez A, Vera-Garcia FJ, De Ste Croix M, Myer GD, Ayala F. Epidemiology of injuries in professional football: a systematic review and meta-analysis. Br J Sports Med. 2020 Jun;54(12):711-718. doi: 10.1136/bjsports-2018-099577. Epub 2019 Jun 6. PMID 31171515
- [Background] Del Coso J, Herrero H, Salinero JJ. Injuries in Spanish female soccer players. J Sport Health Sci. 2018 Apr;7(2):183-190. doi: 10.1016/j.jshs.2016.09.002. Epub 2016 Sep 21. PMID 30356460
- [Background] Schulz KF, Altman DG, Moher, Group C. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar; 340(23): 332.
- [Background] Hermens HJ, Freriks B, Merletti R, Stegeman D, Blok J, Günter R, et al. European Recommendations for Surface ElectroMyoGraphy: Results of the SENIAM Project. Enschede: Roessingh Research and Development; 1999;10 (5): 361-74.